CLINICAL TRIAL: NCT03598036
Title: An Open-Label Dose-Exploration Cohort Study Evaluating the Efficacy and Safety of Voclosporin in Achieving Complete or Partial Remission of Proteinuria in Subjects With Focal Segmental Glomerulosclerosis
Brief Title: Dose-Exploration Evaluating the Efficacy and Safety of Voclosporin in Subjects With Focal Segmental Glomerulosclerosis
Acronym: AURONA™
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUR-VCS-2017-03
Record Dates: First submitted 2018-06-14; First posted 2018-07-26 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2020-06

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: calcineurin inhibitors; Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — voclosporin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Voclosporin (Experimental): Cohort 1:
  Maximum dose of 3 capsules (7.9mg) BID
  Cohort 2
  Dosing to be decided based on the safety from the first 5 or 6 subjects in Cohort 1.
  Interventions: Drug: Voclosporin

INTERVENTIONS:
Drug: Voclosporin — Voclosporin softgel capsules. Up to 10 subjects will be enrolled into Cohort 1 and take up to 3 capsules twice daily (BID).
  The dose of voclosporin for Cohort 2 (at least 10 subjects) will be determined by analysis of efficacy and safety data at Week 12 from the first 5 or 6 subjects in Cohort 1.

SUMMARY:
Evaluating the Efficacy and Safety of Voclosporin in Achieving Complete or Partial Remission of Proteinuria in Subjects with Focal Segmental Glomerulosclerosis

DETAILED DESCRIPTION:
The aim of the current study to assess the efficacy of voclosporin in achieving complete or partial remission of proteinuria after 24 weeks of therapy in subjects with focal segmental glomerulosclerosis (FSGS). As well as to assess the safety and tolerability of voclosporin over 24 weeks in subjects with FSGS.

ELIGIBILITY:
Inclusion Criteria:

1. Primary FSGS diagnosed by renal biopsy.
2. Urine protein creatinine ratio (UPCR) ≥2.0 mg/mg, serum albumin ≤3.2 g/dL and can be immunosuppressant treatment-naïve, or receiving treatment with steroids.
3. Stable proteinuria, renal function, and BP.

Exclusion Criteria:

1. Clinical or histologic evidence of secondary FSGS.
2. Histologic evidence of collapsing variant FSGS.
3. eGFR as calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation of ≤30 mL/minute/1.73 m2 at initial screening assessment or ≤45 mL/minute/1.73 m2 at last qualifying assessment.
4. Currently requiring renal dialysis (hemodialysis or peritoneal dialysis) or expected to require dialysis during the study period.
5. Current or medical history of:

   * Congenital or acquired immunodeficiency.
   * In the opinion of the Investigator, clinically significant drug or alcohol abuse within 2 years prior to screening.
   * Malignancy within 5 years of screening, with the exception of basal and squamous cell carcinomas treated by complete excision.
   * Current or past lymphoproliferative disease or previous total lymphoid irradiation.
   * Severe viral infection within 3 months of screening, or known HIV infection. Severe viral infection is defined as active disease requiring antiviral therapy.
   * Active tuberculosis (TB) or known history of TB/evidence of old TB if not taking prophylaxis with isoniazid.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (20):
  - FSGS Investigative Center, Denver, Colorado
  - FSGS Investigative Center, Winter Park, Florida
  - FSGS Investigative Center, Lawrenceville, Georgia
  - FSGS Investigative Center, Chicago, Illinois
  - FSGS Investigative Center, Iowa City, Iowa
  - FSGS Investigative Center, Louisville, Kentucky
  - FSGS Investigative Center, Shreveport, Louisiana
  - FSGS Investigative Center, Detroit, Michigan
  - FSGS Investigative Center, Minneapolis, Minnesota
  - FSGS Investigative Centre, St Louis, Missouri
  - FSGS Investigative Center, Newark, New Jersey
  - FSGS Investigative Center, New York, New York
  - FSGS Investigative Center, Chapel Hill, North Carolina
  - FSGS Investigative Center, Charlotte, North Carolina
  - FSGS Investigative Center, Columbus, Ohio
  - FSGS Investigative Center, Bethlehem, Pennsylvania
  - FSGS Investigative Center, Dallas, Texas
  - FSGS Investigative Center, El Paso, Texas
  - FSGS Investigative Center, Houston, Texas
  - FSGS Investigative Site, Salt Lake City, Utah
- Dominican Republic (2):
  - FSGS Investigative Centre, Santiago de los Caballeros
  - FSGS Investigative Center, Santo Domingo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ling SY, Huizinga RB, Mayo PR, Larouche R, Freitag DG, Aspeslet LJ, Foster RT. Cytochrome P450 3A and P-glycoprotein drug-drug interactions with voclosporin. Br J Clin Pharmacol. 2014 Jun;77(6):1039-50. doi: 10.1111/bcp.12309. PMID 24330024
- [Background] Ling SY, Huizinga RB, Mayo PR, Freitag DG, Aspeslet LJ, Foster RT. Pharmacokinetics of voclosporin in renal impairment and hepatic impairment. J Clin Pharmacol. 2013 Dec;53(12):1303-12. doi: 10.1002/jcph.166. Epub 2013 Oct 8. PMID 23996158
- [Background] Mayo PR, Huizinga RB, Ling SY, Freitag DG, Aspeslet LJ, Foster RT. Voclosporin food effect and single oral ascending dose pharmacokinetic and pharmacodynamic studies in healthy human subjects. J Clin Pharmacol. 2013 Aug;53(8):819-26. doi: 10.1002/jcph.114. Epub 2013 Jun 4. PMID 23736966
- [Background] Busque S, Cantarovich M, Mulgaonkar S, Gaston R, Gaber AO, Mayo PR, Ling S, Huizinga RB, Meier-Kriesche HU; PROMISE Investigators. The PROMISE study: a phase 2b multicenter study of voclosporin (ISA247) versus tacrolimus in de novo kidney transplantation. Am J Transplant. 2011 Dec;11(12):2675-84. doi: 10.1111/j.1600-6143.2011.03763.x. Epub 2011 Sep 22. PMID 21943027

RESULTS

PARTICIPANT FLOW:
Groups:
- Voclosporin Cohort 1: Cohort 1:
  Maximum dose of 3 capsules voclosporin (23.7 mg total) twice daily
- Voclosporin Cohort 2: Trial ended prematurely before any patients were enrolled into Cohort 2
  Cohort 2:
  When Cohort 1 have completed 12 weeks of treatment with voclosporin, the top line efficacy and safety data will be analyzed to determine the dose level for Cohort 2. The selected dose may be higher or lower than 23.7 mg twice daily.
  The maximum dose possible for Cohort 2 will be 39.5 mg (5 capsules) twice daily.
Period: Overall Study
Arm/Group | Voclosporin Cohort 1 | Voclosporin Cohort 2
Started | 5 | 0 (Trial ended prematurely before any patients were enrolled into Cohort 2)
Week 1: 7.9 mg Twice Daily | 5 | 0
Week 2: 15.9 mg Twice Daily | 5 | 0
Weeks 3 - 24: 23.7 mg Twice Daily | 5 (1 subject withdrew at Week 12) | 0
Completed | 4 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Trial ended prematurely before any patients were enrolled into Cohort 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Voclosporin Cohort 1 | Voclosporin Cohort 2 | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (20.71) |  | 36.2 (20.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 3 |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 |  | 2
  Not Hispanic or Latino | 3 |  | 3
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3
  Dominican Republic | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Remission of Proteinuria
Description: Complete remission OR Partial remission
Time Frame: 24 weeks
Population: Due to difficulties enrolling appropriate Focal Segmental Glomerulosclerosis (FSGS) patients, Aurinia terminated the clinical trial early. Focal Segmental Glomerulosclerosis (FSGS) is a rare disease with an estimated 40,000 adult patients in the USA. Only five subjects were enrolled into the clinical trial. The primary and secondary endpoints were not assessed due to insufficient data collected
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

2. Secondary Outcome: Proportion of Subjects With Complete Remission or Partial Remission of Proteinuria
Description: Complete remission or partial remission of proteinuria
Time Frame: Weeks 8 and 12
Population: as for outcome 1
Groups:
- Voclosporin Cohort 1: Cohort 1:
  Maximum dose of 3 capsules voclosporin (23.7mg total) twice daily
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Subjects With Complete Remission of Proteinuria
Description: Complete remission of proteinuria
Time Frame: Weeks 8, 12, and 24
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

4. Secondary Outcome: Proportion of Subjects With Reduction of Proteinuria
Description: Reduction of proteinuria
Time Frame: Weeks 8, 12, and 24
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

5. Secondary Outcome: Proportion of Subjects With Partial Remission of Proteinuria
Description: Partial remission of proteinuria
Time Frame: Weeks 8, 12, and 24
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to First Occurrence of Complete or Partial Remission of Proteinuria
Description: Complete OR partial remission of proteinuria
Time Frame: Up to 26 weeks
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

7. Secondary Outcome: Time to First Occurrence of Complete Remission of Proteinuria
Description: Complete remission of proteinuria
Time Frame: Up to 26 weeks
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

8. Secondary Outcome: Time to First Occurrence of Partial Remission of Proteinuria
Description: Partial remission of proteinuria
Time Frame: Up to 26 weeks
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

9. Secondary Outcome: Time to First Occurrence of 50% Reduction in Urine Protein Creatinine Ratio (UPCR) From Baseline
Description: 50% reduction in Urine Protein Creatinine Ratio (UPCR) from baseline
Time Frame: Up to 26 weeks
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

10. Secondary Outcome: Duration of Reduced Urine Protein Creatinine Ratio (UPCR)
Description: Duration of reduced Urine Protein Creatinine Ratio (UPCR)
Time Frame: Up to 26 weeks
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline in Urine Protein Creatinine Ratio (UPCR)
Description: Change from baseline in Urine Protein Creatinine Ratio (UPCR)
Time Frame: Weeks 2,4,8,12,18,24
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

12. Secondary Outcome: Proportion of Subjects With a Confirmed Decrease From Baseline in Estimated Glomerular Filtration Rate (eGFR)
Description: Utilizing the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula
Time Frame: Weeks 2,4,8,12,18,24
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

13. Secondary Outcome: Proportion of Subjects With a Confirmed Increase in Estimated Glomerular Filtration Rate (eGFR)
Description: Increase in Estimated Glomerular Filtration Rate (eGFR)
Time Frame: Week 24 to Week 26
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

14. Secondary Outcome: Change in Urine Protein Creatinine Ratio (UPCR)
Description: Change in Urine Protein Creatinine Ratio (UPCR)
Time Frame: Week 24 and Week 26
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

15. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR)
Description: Change in estimated Glomerular Filtration Rate (eGFR)
Time Frame: Week 24 and Week 26
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

16. Secondary Outcome: Change From Baseline in Serum Creatinine, Serum Albumin and Estimate Glomerular Filtration Rate (eGFR)
Description: Change from baseline in serum creatinine, serum albumin and estimate Glomerular Filtration Rate (eGFR)
Time Frame: Weeks 2,4,8,12,18,24
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

17. Secondary Outcome: Quality of Life Assessments
Description: Mean change in Patient Reported Outcome Measurement Information System (PROMIS) measures
Time Frame: Week 24
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

18. Secondary Outcome: Quality of Life Assessments
Description: Change from baseline in Kidney Disease Quality of Life-Short Form (KDQOL-SF)
Time Frame: Week 24
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

19. Secondary Outcome: Safety and Tolerability (Treatment-Emergent Adverse Events)
Description: Incidence and number of treatment-emergent adverse events
Time Frame: 24 weeks
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

20. Secondary Outcome: Renal Biopsy
Description: Descriptive analyses of changes in histopathology will be evaluated in post treatment renal biopsies in a subset of patients
Time Frame: 24 weeks
Population: as for outcome 1
Arm/Group | Voclosporin Cohort 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Week 26
Description: Trial ended prematurely before any patients were enrolled into Cohort 2
Groups:
- Voclosporin Cohort 1: Week 1: Cohort 1: Week 1 7.9 mg twice daily
- Voclosporin Cohort 1: Week 2: Cohort 1: Week 2 15.9 mg twice daily
- Voclosporin Cohort 1: Weeks 3-24: Cohort 1: Weeks 3-24 23.7 mg twice daily
Arm/Group | Voclosporin Cohort 1: Week 1 | Voclosporin Cohort 1: Week 2 | Voclosporin Cohort 1: Weeks 3-24 | Voclosporin Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 1/5 | 0/0
Other Adverse Events (participants affected / at risk) | 2/5 | 0/5 | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voclosporin Cohort 1: Week 1 (N=5) | Voclosporin Cohort 1: Week 2 (N=5) | Voclosporin Cohort 1: Weeks 3-24 (N=5) | Voclosporin Cohort 2 (N=0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voclosporin Cohort 1: Week 1 (N=5) | Voclosporin Cohort 1: Week 2 (N=5) | Voclosporin Cohort 1: Weeks 3-24 (N=5) | Voclosporin Cohort 2 (N=0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | NA
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 3 (3) | NA
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | NA
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2) | NA
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | NA
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | NA
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | NA
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
Due to difficulties enrolling appropriate Focal Segmental Glomerulosclerosis (FSGS) patients, Aurinia terminated the clinical trial early. Focal Segmental Glomerulosclerosis (FSGS) is a rare disease with an estimated 40,000 adult patients in the USA. Only five subjects were enrolled into the clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Protocol v1.0 (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT03598036/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Protocol v2.0 (Amendment 1) (2018-11-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT03598036/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: Protocol v3.0 (Amendment 2) (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT03598036/Prot_SAP_002.pdf
  • Study Protocol and Statistical Analysis Plan: Protocol v4.0 (Amendment 3) (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03598036/Prot_SAP_003.pdf